CLINICAL TRIAL: NCT04372927
Title: Adaptive-Dose to Mediastinum With Immunotherapy (Durvalumab MEDI4736) and Radiation in Locally-Advanced Non-Small Cell Lung Cancer
Brief Title: ADMIRAL Trial: Adaptive Mediastinal Radiation With Chemo-Immunotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jing Zeng, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1007190; NCI-2020-02417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10459 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Etoposide; Radiation Dose Hypofractionation; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, durvalumab, radiation therapy) (Experimental): Patients with squamous cell cancer receive standard of care chemotherapy consisting of cisplatin on days 1, 8, 29, and 36, and etoposide on days 1-5 and 29-33. Cycles repeat every 4 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with non-squamous cell cancer receive standard of care chemotherapy consisting of cisplatin and pemetrexed on days 1, 22, and 43. Cycles repeat every 3 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. All patients receive durvalumab IV over 1 hour Q4W. Radiation to the primary tumor will be given over 8-15 fractions during weeks 1-3 of chemotherapy. For patients who have residual disease in the mediastinal lymph nodes at week 9, radiation will be given to the lymph nodes starting week 11. Durvalumab is given for 2 years after completion of radiation in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Biological: Durvalumab; Drug: Etoposide; Radiation: Hypofractionated Radiation Therapy; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736; 1428935-60-7
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy

SUMMARY:
This phase II trial studies two questions in patients with stage III NSCLC: 1) does it improve cancer control to add the drug Durvalumab, a type of immunotherapy, earlier in the treatment course; and 2) by intensifying treatment with durvalumab, is it possible to avoid mediastinal radiation to decrease side effects, without decreasing cancer control?

DETAILED DESCRIPTION:
OUTLINE:

Patients will receive platinum doublet chemotherapy per standard of care with durvalumab for 8 weeks, concurrent with a short course of radiation to the primary lung tumor. Patients will then undergo repeat evaluation of the mediastinal lymph nodes. If there is no cancer in the lymph nodes, patients will receive 2 years of adjuvant durvalumab. If there is still cancer in the lymph nodes, patients will receive 6 weeks of radiation to the mediastinal lymph nodes, and 2 years of adjuvant durvalumab.

After the completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-small cell lung cancer (NSCLC)
* Stage III NSCLC according to American Joint Committee on Cancer (AJCC) staging version (v)8
* At least one mediastinal site of disease that is discontiguous from all other visible sites of disease and can be excluded from primary tumor site radiation (i.e. at least 10 mm separation between tumors)
* A maximum of 20 patients with bulky mediastinal disease will be allowed on this trial, defined as at least one contiguous mediastinal mass with minimum diameter > 2 cm, that is not contiguous with the primary tumor (and therefore would not be irradiated during radiation to the primary tumor)
* No surgery for lung cancer for at least 3 years
* No other malignancies for at least 3 years, excluding low grade or non-invasive malignancies such as skin cancers, prostate cancers, and ductal breast carcinoma in situ (DCIS)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Age >= 18 years at time of study entry
* Life expectancy of >= at least 3 months
* Body weight > 30 kg
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) 1.5 (or 1.0) x (>= 1500 per mm^3)
* Platelet count >= 100,000 per mm^3
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine transferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x upper limit of normal (ULN)
* Measured creatinine clearance (CL) > 60 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Prior anti-CTLA-4, PD-1 or PD-L1 antibodies including durvalumab
* Prior chemotherapy in the past 3 years from consent
* Any unresolved toxicity National Cancer Institute (NCI) CTCAE grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
* Prior thoracic radiation that would preclude curative-intent radiation dose as outlined in this study
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product (IP). Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Progression-free Survival Rate (PFS)
Description: Will be evaluated using the method of Kaplan-Meier. Confidence intervals for median times will be determined using the Brookmeyer-Crowley method. Confidence intervals around landmark times will be determined using Greenwood's formula for the variance and based on a log-log transformation applied on the survival function. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as response. Means and/or medians will be calculated for continuous outcomes. Confidence bounds will be provided for means and quartiles and ranges for median values. All confidence bounds will be presented as 95% bounds.
Time Frame: Study enrollment to disease progression or death, whichever occurs first, for up to 1 year
Population: No patient was alive at 1 year.
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency and Severity of Pneumonitis
Description: The primary toxicity of interest is grade 3 or higher pneumonitis. The incidence of grade 3 or worse pneumonitis attributable to treatment will be evaluated and compared against the PACIFIC trial results. All toxicities of all grades will be monitored on study and reported. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as toxicity.
Time Frame: Through study completion (up to 4 months)
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 1
participants | 1

3. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 1
Time Frame: From study registration to death due to any cause
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 1
months | 4 (NA) — Standard Deviation is not calculable for 1 participant

4. Secondary Outcome: Response Rate
Description: as for outcome 1
Time Frame: Through study completion (up to 4 months)
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 1
participants | 0

5. Secondary Outcome: Frequency of Adverse Events
Description: Frequency and severity of toxicities will be graded with Common Terminology Criteria for Adverse Events (CTCAE), version 5. Toxicities will be summarized as the proportion of patients with such toxicities, in addition to total number of toxicities (allowing for multiple toxicities within a patient) among all patients. All toxicities of all grades will be monitored on study and reported. Binary proportions will be calculated with associated confidence intervals for binary outcomes, such as toxicity.
Time Frame: Through study completion (up to 4 months)
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 4 months
Description: CTCAE v5
Arm/Group | Treatment (Chemotherapy, Durvalumab, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Durvalumab, Radiation Therapy) (N=1)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Durvalumab, Radiation Therapy) (N=1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
We enrolled one participant, then trial closed due to poor accrual. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04372927/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT04372927/ICF_000.pdf